CLINICAL TRIAL: NCT02711358
Title: Rectal Indomethacin Use in Pain Relief During Intrauterine Device Insertion: A Randomized Controlled Trial
Brief Title: Indomethacin Use in Pain Relief During Intrauterine Device Insertion
Acronym: INDO-IUD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: INDO
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Family Planning

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- indomethacin (Experimental): indomethacin suppositories
  Interventions: Drug: indomethacin suppositories
- placebo (Placebo Comparator): placebo suppositories
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: indomethacin suppositories — The patients will be instructed to self-administer a single rectal dose of 50 mg indomethacin 30 min before the scheduled time of the procedure
  Arms: indomethacin
Drug: placebo — The patient swill be instructed to self-administer a single rectal dose of placebo 30 min before the scheduled time of the procedure
  Arms: placebo

SUMMARY:
The aim of the investigators study is to test the analgesic effect of rectal indomethacin during Intrauterine device insertion.

ELIGIBILITY:
Inclusion Criteria:

* Women not taken analgesics or anxiolytics in the 24 hours prior insertion
* Women not taken misoprostol prior to intrauterine device insertion
* Women who will accept to participate in the study

Exclusion Criteria:

* Any contraindication to intrauterine device placement

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Mean pain score during IUD insertion | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided